CLINICAL TRIAL: NCT01970410
Title: MAIN STUDY: Switching Relapsing Multiple Sclerosis Patients Treated With Natalizumab at Risk for Progressive Multifocal Leukoencephalopathy to Teriflunomide: Is This Safe and Effective? SUB-STUDY: Analysis of JCV Antibody Index in MS Patients Treated With Teriflunomide
Brief Title: MAIN STUDY: SWITCH SUB-STUDY: SWITCH-JCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Multiple Sclerosis Center of Northeastern New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWITCH-001
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
Keywords: teriflunomide; natalizumab; relapsing multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Teriflunomide (Experimental): Teriflunomide 14 mg oral teriflunomide daily
  Interventions: Drug: teriflunomide

INTERVENTIONS:
Drug: teriflunomide — 14 mg oral teriflunomide daily
  Other Names: Aubagio

SUMMARY:
MAIN STUDY: The purpose of this study is to determine if teriflunomide will be safe and effective to prevent relapses in patients with relapsing types of MS when switching from natalizumab to teriflunomide in patients at risk for PML. This is a two center interventional study of patients who have had 12 or more continuous infusions of natalizumab , who are anti-JCV-ab positive, and who had been free of clinical relapses during prior 12 months of natalizumab therapy who will be switching to teriflunomide.

SUB-STUDY: To study the number of patients experiencing a reduction in the anti-JCV antibody Index value in patients who had received at least one dose of teriflunomide during participation in the SWITCH protocol (main study).

DETAILED DESCRIPTION:
MAIN STUDY: Teriflunomide (TFM) is the primary metabolite of leflunomide, which is marketed worldwide for the treatment of rheumatoid arthritis. Teriflunomide inhibits dihydroorotate dehydrogenase( DHODH), the forth enzyme in the de novo synthesis pathway of pyrimidines. Activated T-lymphocytes utilize both the de novo pyrimidine and salvage pathways of pyrimidines ribonucleotide synthesis.After mitogen stimulation, teriflunomide inhibits in vitro T cell proliferation, DNA and RNA synthesis and expression of cell surface and nuclear antigens that are directly involved in T-cell activation and proliferation.

Natalizumab (NTZ) is a FDA approved treatment for relapsing-forms of multiple sclerosis (MS) with pivotal studies showing an annualized relapse-rate (ARR) reduction of 68%, a reduction of new Gadolinium "enhancing" (Gd+) lesions by 92% and a reduction of disability of 42% compared to placebo. NTZ is highly effective in controlling MS but the risk of developing progressive multifocal leukoencephalopathy (PML) increases with the duration of the use of natalizumab. It can have a serious and life threatening complication in about 1 in 500 to 1 in 250 patients who have had more that 18 infusions due PML and who have a detected antibody (Ab) for the JC virus. The risk of PML is much greater in patients who have had prior immunosuppressive (IS) treatment. The combination of detected anti-JCV Ab , duration of NTZ treatment of greater than 24 months and prior IS increases the risk of development PML to an incidence of 11 per 1000 treated patients. So there is a need to have an alternative MS disease modifying treatment (DMT) to use for patients at risk to develop PML from NTZ treatment that might be sufficiently effective for MS so as not to have the patients' MS worsen while lowering or eliminating the risk of PML.

SUB-STUDY: John Cunningham virus (JCV) is the responsible organism for the development of progressive multifocal encephalopathy (PML). Multiple sclerosis (MS) patients treated with natalizumab (NTZ), who have evidence of exposure to JCV have a significantly elevated risk, as high as 12/1000 patients, of developing PML, necessitating the elective transition of patients off NTZ.

JCV is a member of the polyoma virus family, and closely related to BK virus. BK virus has been found to be a significant threat to destroy transplanted kidneys and there is growing evidence that treatment with leflunomide, the pro-drug of teriflunomide (TFM) clears BKV from the kidney.

Main study assessed the clinical efficacy of TFM in MS patients transitioned off NTZ solely because they have evidence of exposure to JCV, as determined by the presence of serum anti-JCV immunoglobulin G (IgG). Previous work by other investigators has demonstrated a close correlation between positive anti-JCV antibody titers and the presence of active JCV infection.

There is evidence that JCV is closely related to its fellow polyoma virus BKV, and that BKV is cleared by treatment with the TFM pro-drug leflunomide, we propose to determine if treatment of the JCV antibody positive patients currently enrolled in the approved protocol results in reduction in, or reversion to negative, of the anti-JCV antibody titer as measured by the JCV antibody Index, a commercially available assay which is used internationally as the standard for evidence of JCV exposure in NTZ-treated patients.

ELIGIBILITY:
MAIN STUDY

Inclusion Criteria:

* Male and female patients, age 21 to 60 with relapsing forms of MS, treated with natalizumab for 12 consecutive months or longer with anti-JCV Ab positive during that time period.
* Able to understand and sign Informed Consent Document.
* Stable disease during treatment with natalizumab. No clinical relapses for at least 12 months.
* Stable MRI on follow-up MRI scans for prior 12 months without evidence of new or enlarging T-2 hyperintensities or Gd+ lesions.
* No clinical evidence by imaging or cerebrospinal fluid (CSF) for PML.
* No evidence of significant cognitive limitation or psychiatric disorder.
* Expanded Disability Status Scale (EDSS) of 1.0 to 6.0 inclusive.

Exclusion Criteria:

* Any mental condition of such that patient is unable to understand the nature, scope and possible consequences of the study.
* Patients that are known HIV positive.
* Patients with a known history of hepatitis.
* Known history of active tuberculosis not adequately treated, or a positive ppd skin test or positive quantiferon gold.
* Any persistent or severe infection.
* Any malignancy within 5 years, except for Basal or Squamous cell skin lesions, which have been surgically excised, with no evidence of metastasis.
* Clinically relevant or unstable cardiovascular, neurological (i.e. progressive weakness, increasing hypesthesia), endocrine, or other major systemic diseases.
* History of drug or alcohol abuse within the past year.
* Any significant depression or psychiatric disease (BDI II greater than 25) within the past year.
* Any significant lab abnormality as deemed by the investigator including but not limited to the following:

  1. Hypoproteinemia with serum albumin < 3.0g/dl.
  2. Serum creatinine >133umol/L (or >1.5 mg/dl)
  3. Hematocrit <24% and/or
  4. Absolute white blood cell count < 4,000 cells/mm3 (µl) and/or
  5. Platelet Count <150,000 cells/mm3 (µl) and /or
  6. Absolute neutrophil < 1,500 cells/mm3 (µl)
  7. Liver function impairment or persisting elevations of serum glutamate pyruvate transaminase (SGPT)/ Alanine transaminase (ALT), serum glutamate oxaloacetate transaminase (SGOT)/ aspartate aminotransferase (AST), or direct bilirubin greater than 1.5 fold the upper limit of normal.
* Any confounding illness or other diseases of the spine or bone that would impair evaluation of the patient or treatment effects.
* Any clinical, CSF or MRI evidence for PML.
* Prior treatment with immunosuppressive drugs except for past use of intravenous steroids to treat MS relapses.
* Pregnant or breast feeding women.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or are unwilling or unable to be tested for pregnancy.
* In the conception of a child during the course of the trial.
* Known history of hypersensitivity to teriflunomide or leflunomide.
* Persisting elevations (confirmed by retest) of serum amylase or lipase greater than 2-fold the upper limit of normal.
* Known history of chronic pancreatic disease or pancreatitis.
* Prior use within 4 weeks before randomization or concomitant use of phenytoin, warfarin, tolbutamide, cholestyramine, or products containing St. John's Wort

SUB-STUDY

Eligibility Criteria for JCV sub-study:

* Must have been enrolled in the SWITCH protocol and received at least 1 dose of 14mg TFM during the study period.
* Must be willing to sign written, informed consent for this JCV sub-study and follow protocol requirements.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2013-10; Primary Completion 2021-04-30 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, MD, Study Director — Multiple Sclerosis Center of Northeastern New York; Stanley Cohan, MD, Ph. D, Principal Investigator — Providence Multiple Sclerosis Center
Locations (3):
- United States (3):
  - Phoenix Neurological Associates, Ltd, Phoenix, Arizona
  - Multiple Sclerosis Center of Northeastern New York, Latham, New York
  - Providence Multiple Sclerosis Center, Portland, Oregon

REFERENCES:
- [Background] Gold R, Wolinsky JS. Pathophysiology of multiple sclerosis and the place of teriflunomide. Acta Neurol Scand. 2011 Aug;124(2):75-84. doi: 10.1111/j.1600-0404.2010.01444.x. Epub 2010 Sep 29. PMID 20880295
- [Background] Fox RI, Herrmann ML, Frangou CG, Wahl GM, Morris RE, Strand V, Kirschbaum BJ. Mechanism of action for leflunomide in rheumatoid arthritis. Clin Immunol. 1999 Dec;93(3):198-208. doi: 10.1006/clim.1999.4777. PMID 10600330
- [Background] Ruckemann K, Fairbanks LD, Carrey EA, Hawrylowicz CM, Richards DF, Kirschbaum B, Simmonds HA. Leflunomide inhibits pyrimidine de novo synthesis in mitogen-stimulated T-lymphocytes from healthy humans. J Biol Chem. 1998 Aug 21;273(34):21682-91. doi: 10.1074/jbc.273.34.21682. PMID 9705303
- [Background] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Background] Gorelik L, Lerner M, Bixler S, Crossman M, Schlain B, Simon K, Pace A, Cheung A, Chen LL, Berman M, Zein F, Wilson E, Yednock T, Sandrock A, Goelz SE, Subramanyam M. Anti-JC virus antibodies: implications for PML risk stratification. Ann Neurol. 2010 Sep;68(3):295-303. doi: 10.1002/ana.22128. PMID 20737510
- [Background] Bloomgren G, Richman S, Hotermans C, Subramanyam M, Goelz S, Natarajan A, Lee S, Plavina T, Scanlon JV, Sandrock A, Bozic C. Risk of natalizumab-associated progressive multifocal leukoencephalopathy. N Engl J Med. 2012 May 17;366(20):1870-80. doi: 10.1056/NEJMoa1107829. PMID 22591293
- [Background] Miravalle A, Jensen R, Kinkel RP. Immune reconstitution inflammatory syndrome in patients with multiple sclerosis following cessation of natalizumab therapy. Arch Neurol. 2011 Feb;68(2):186-91. doi: 10.1001/archneurol.2010.257. Epub 2010 Oct 11. PMID 20937940
- [Background] Stuve O, Cravens PD, Frohman EM, Phillips JT, Remington GM, von Geldern G, Cepok S, Singh MP, Tervaert JW, De Baets M, MacManus D, Miller DH, Radu EW, Cameron EM, Monson NL, Zhang S, Kim R, Hemmer B, Racke MK. Immunologic, clinical, and radiologic status 14 months after cessation of natalizumab therapy. Neurology. 2009 Feb 3;72(5):396-401. doi: 10.1212/01.wnl.0000327341.89587.76. Epub 2008 Nov 5. PMID 18987352
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Result] Cohan SL, Edwards K, Lucas L, Gervasi-Follmar T, O'Connor J, Siuta J, Kamath V, Garten L, Chen C, Thomas J, Smoot K, Kresa-Reahl K, Spinelli KJ. Reducing return of disease activity in patients with relapsing multiple sclerosis transitioned from natalizumab to teriflunomide: 12-month interim results of teriflunomide therapy. Mult Scler J Exp Transl Clin. 2019 Jan 16;5(1):2055217318824618. doi: 10.1177/2055217318824618. eCollection 2019 Jan-Mar. PMID 30729028
- [Result] Cohan S, Gervasi-Follmar T, Kamath A, Kamath V, Chen C, Smoot K, Baraban E, Edwards K. The results of a 24-month controlled, prospective study of relapsing multiple sclerosis patients at risk for progressive multifocal encephalopathy, who switched from prolonged use of natalizumab to teriflunomide. Mult Scler J Exp Transl Clin. 2021 Dec 16;7(4):20552173211066588. doi: 10.1177/20552173211066588. eCollection 2021 Oct. PMID 34950502

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriflunomide: Oral teriflunomide treatment 14 mg a day 28 ± 7 days after last natalizumab infusion.
Period: Main Study
Arm/Group | Teriflunomide
Started | 55
Baseline Procedures | 55
Completed | 28
Not Completed | 27
Period: Sub-Study
Arm/Group | Teriflunomide
Started | 41
Completed | 36
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Main study participants.
Arm/Group | Teriflunomide
Number analyzed (Participants) | 55
Age, Continuous [Median (Inter-Quartile Range); unit: Years]
  Main Study | 47.0 [40.7 to 56.3]
Age, Continuous [Median (Standard Deviation); unit: Years] — Age, continuous for Sub-study. Population: Row population differs from the Overall as there was a sub study to the main study. Of the 55 participants who partook in the main study, 36 participated in the sub-study.
  Years
    Sub-Study: number analyzed (Participants) | 36
    Sub-Study | 49.13 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Main Study: Female | 42
  Main Study: Male | 13
Sex: Female, Male [Count of Participants; unit: Participants] — Sex: Female, Male for sub-study. Population: Row population differs from the Overall as there was a sub study to the main study. Of the 55 participants who partook in the main study, 36 participated in the sub-study.
  Participants
    Sub-Study: number analyzed (Participants) | 36
    Sub-Study: Female | 28
    Sub-Study: Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Main Study: American Indian or Alaska Native | 0
  Main Study: Asian | 0
  Main Study: Native Hawaiian or Other Pacific Islander | 0
  Main Study: Black or African American | 2
  Main Study: White | 53
  Main Study: More than one race | 0
  Main Study: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race for sub-study. Population: Row population differs from the Overall as there was a sub study to the main study. Of the 55 participants who partook in the main study, 36 participated in the sub-study.
  Participants
    Sub-Study: number analyzed (Participants) | 36
    Sub-Study: American Indian or Alaska Native | 0
    Sub-Study: Asian | 0
    Sub-Study: Native Hawaiian or Other Pacific Islander | 0
    Sub-Study: Black or African American | 1
    Sub-Study: White | 35
    Sub-Study: More than one race | 0
    Sub-Study: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Region of Enrollment for MAIN study.
  participants
    United States | 55
Region of Enrollment [Number; unit: participants] — Region of enrollment number for Sub-study. Population: Row population differs from the Overall as there was a sub study to the main study. Of the 55 participants who partook in the main study, 36 participated in the sub-study.
  participants
    United States: number analyzed (Participants) | 36
    United States | 36
Duration of prior Natalizumab in years [Median (Inter-Quartile Range); unit: Years] — Duration of prior Natalizumab in years for MAIN study.
  Years | 2.8 [1.5 to 5.3]
Duration of prior NTZ in years [Median (Inter-Quartile Range); unit: Years] — Duration of prior NTZ in years for SUB-study. Population: Row population differs from the Overall as there was a sub study to the main study. Of the 55 participants who partook in the main study, 36 participated in the sub-study.
  Years
    number analyzed (Participants) | 36
    (all) | 3.71 [1.38 to 5.09]

OUTCOME MEASURES:

1. Primary Outcome: MAIN STUDY: Number of Participants Relapse Free at 24 Months
Description: Number of patients relapses free by month 24.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide
Number analyzed (Participants) | 55
Participants | 25

2. Secondary Outcome: MAIN STUDY: Time to Return of Radiological Evidence of Multiple Sclerosis Activity With New Gadolinium "Enhancing" (Gd+) Lesions on Cranial MRI.
Description: Mean time to first Gadolinium "enhancing" (GAD+) lesion in months.
Time Frame: 24 months
Measure: Mean (Standard Error); unit: Months
Arm/Group | Teriflunomide
Number analyzed (Participants) | 55
Months | 19.6 (1.1)

3. Secondary Outcome: MAIN STUDY: Expanded Disability Status Scale (EDSS) Sustained Progression for 3 Months as Measured by at Least 0.5 Increase From Baseline or 1 in Any EDSS Set Score
Description: Mean time to 3-month sustained disability worsening (SDW) in months. SDW is defined as an increase of ≥ 1 point for patients with EDSS of 1.0-5.0, and ≥ 0.5 points for patients with an EDSS of 5.5-6.0, sustained for 3 months. Patients with ≥ 1 point increase in EDSS in whom a second measure was not obtained 3 months later were not included as SDW.
Time Frame: 24 months
Measure: Mean (Standard Error); unit: Months
Arm/Group | Teriflunomide
Number analyzed (Participants) | 55
Months | 22 (0.7)

4. Secondary Outcome: MAIN STUDY: Mean Time to New T2 or Enlarging T2 Hyperintensities on Monthly Sentinel Brain MRIs
Description: Mean time of new T2 or enlarging T2 Lesions
Time Frame: 24 months
Measure: Mean (Standard Error); unit: Months
Arm/Group | Teriflunomide
Number analyzed (Participants) | 55
Months | 19.2 (1.1)

5. Post Hoc Outcome: SUB-STUDY: Number of Patients With a Reduction of Anti-JCV Antibody Index (AJAI)
Description: Number of patients with a >= 20% reduction of AJAI.
  The AJAI serostatus categories used in the study were negative (<0.2), positive (0.41-0.89) and high positive (≥0.90). The 0.2-0.4 range is frequently reported as indeterminate. We defined a change of 20% or greater as a meaningful increase or decrease in the AJAI.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Anti-JCV Antibody Status (Sub-Study): Number of patients with a reduction in the anti-JCV antibody Index value who received Teriflunomide,14 mg oral teriflunomide daily.
Arm/Group | Anti-JCV Antibody Status (Sub-Study)
Number analyzed (Participants) | 36
Participants | 20

ADVERSE EVENTS:
Time Frame: 24 months for the main study and 5 days after blood draw for the sub-study
Groups:
- MAIN STUDY: Teriflunomide: Oral teriflunomide treatment 14 mg a day 28 ± 7 days after last natalizumab infusion.
- SUB-STUDY: Anti- John Cunningham Virus (JCV) Antibody Status: Analysis of JCV Antibody Index in MS Patients treated with teriflunomide.
Arm/Group | MAIN STUDY: Teriflunomide | SUB-STUDY: Anti- John Cunningham Virus (JCV) Antibody Status
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/36
Serious Adverse Events (participants affected / at risk) | 5/55 | 0/36
Other Adverse Events (participants affected / at risk) | 47/55 | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAIN STUDY: Teriflunomide (N=55) | SUB-STUDY: Anti- John Cunningham Virus (JCV) Antibody Status (N=36)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrenous appendicitis, ruptured (Infections and infestations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Right pneumothorax (Infections and infestations) | 1 (1) | 0 (0)
Squamous cell carcinoma, left ankle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subfalcial herniation (Nervous system disorders) | 1 (1) | 0 (0)
Obstructive hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAIN STUDY: Teriflunomide (N=55) | SUB-STUDY: Anti- John Cunningham Virus (JCV) Antibody Status (N=36)
Hair Thinning/ loss (Skin and subcutaneous tissue disorders) | 20 (20) | 0 (0)
Diarrhea /loose stool (Gastrointestinal disorders) | 18 (18) | 0 (0)
Headache (Nervous system disorders) | 12 (12) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 11 (11) | 0 (0)
Vertigo/balance difficulty/dizziness (Nervous system disorders) | 11 (11) | 0 (0)
Fatigue (Nervous system disorders) | 10 (10) | 0 (0)
Tingling/paresthesia (Nervous system disorders) | 10 (10) | 0 (0)
Upper respiratory infection (Infections and infestations) | 10 (10) | 0 (0)
Cognitive changes (Nervous system disorders) | 8 (8) | 0 (0)
Elevated transaminase (Blood and lymphatic system disorders) | 8 (8) | 0 (0)
Extremity joint pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Other infections (Infections and infestations) | 8 (8) | 0 (0)
Sensory decrease/disturbance (Nervous system disorders) | 8 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 0 (0)
Depression (Psychiatric disorders) | 8 (8) | 0 (0)
Rashes/eczema (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Abdominal pain/discomfort (Gastrointestinal disorders) | 6 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 0 (0)
Ophthalmic changes (Eye disorders) | 6 (6) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 5 (5) | 0 (0)
Heartburn (Gastrointestinal disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)
Stiffness/spasticity (Nervous system disorders) | 5 (5) | 0 (0)
Migraine (Nervous system disorders) | 5 (5) | 0 (0)
Skin irritation secondary to multiple tries to perform draw and bruising at site of blood draw (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Sub Study (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT01970410/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Main Study (2015-02-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT01970410/Prot_SAP_001.pdf
  • Informed Consent Form: Sub Study (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT01970410/ICF_002.pdf
  • Informed Consent Form: Main study (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT01970410/ICF_003.pdf